CLINICAL TRIAL: NCT03227887
Title: Evaluation of the Link Between the Characteristics of Oral Physiology and Formation of the Food Bolus During the Consumption of Cereal Products in Elderly People Via a Modelling Approach.
Brief Title: Evaluate the Link Between the Characteristics of Oral Physiology and the Formation of the Food Bolus During the Consumption of Cereal Products in Elderly People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: VVW Alimassens cereales
Record Dates: First submitted 2017-06-26; First posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Old Person

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Good chewing ability (Active Comparator)
  Interventions: Other: Two samples of saliva; Other: Chewing behaviour; Other: Study of the food bolus; Other: Mouthfeel
- Impaired chewing ability (Experimental)
  Interventions: Other: Two samples of saliva; Other: Chewing behaviour; Other: Study of the food bolus; Other: Mouthfeel

INTERVENTIONS:
Other: Two samples of saliva — 1. Without stimulation : the 1st will be used to measure the flow of naturally secreted saliva
  2. With stimulation: The 2nd will be used to measure the flow and viscosity of the saliva secreted after stimulation
Other: Chewing behaviour — Measure the time taken by the subjects to chew the food and the number of bites they use before swallowing The test will be done twice.
Other: Study of the food bolus — 2 tests:
  1. Evaluate using a compression test the structure of each bolus to determine their degree of destructuration over time Measure the quantity of the saliva incorporated
  2. The bolus will be analysed visually
Other: Mouthfeel — Describe the mouthfeel by answering a paper questionnaire after consumption of the cereal products

SUMMARY:
The aim of this study is to understand how foods such as Sponge cake or Brioche are broken down in the mouth. More specifically, investigators wish to evaluate the link between oral physiology (salivation and mastication) and (i) formation of the food bolus during the consumption of Sponge cake or Brioche, that is to say the way in which the food is broken down to be swallowed (ii) mouthfeel during the consumption of Sponge cake or Brioche, meaning the sensations that participant feel when they eat these products.

The study will take place at the INRA in Dijon during 7 one-hour sessions spread over 3 months. The first session will allow us to characterise the chewing behaviour of the subjects and their salivation, and will enable us to train them in the instructions for the following sessions. The 6 other sessions will allow us to study the structure of the food bolus while being formed and the mouthfeel of the foods in the project.

In the first session:

* Two samples of saliva will be taken
* A video will be made of subjects eating Sponge cake or Brioche
* Subjects will be trained in exercises for the following sessions - this will consist in chewing the study foods and spitting them out on the experimenter's signal.

During the 6 other sessions, subjects will be asked to:

* Chew one of the study foods and spit it out on the signal of the experimenter.
* Evaluate the mouthfeel while eating Sponge cake or Brioche by answering different questions. This test will be done during 4 of the 6 sessions.

ELIGIBILITY:
Inclusion Criteria:

* persons who have provided written consent
* Age ≥ 65 years old
* Persons living at home
* Persons who can travel independently

Exclusion Criteria:

* Adults under guardianship
* Persons without health insurance cover
* Persons in hospital
* Persons in institutions
* Persons whose Mini-Mental State Examination (MMSE) is < 24
* Persons requiring enteral or parenteral nutrition
* Persons who in the previous 12 months received € 4500 for taking part in clinical trials, including the present study
* Persons in a period of exclusion of a previous study
* Food allergies (cereal products in particular)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-06-06 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Duration of chewing during consumption of cereal products | At baseline
Frequency of chewing during consumption of cereal products | At baseline
Rheology test | Up to 3 months
Calculation of insalivation rates | Up to 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France